CLINICAL TRIAL: NCT02518542
Title: Per Oral Endoscopic Myotomy (POEM) and Prolonged Dilatation (PRD) as Additional Endoscopic Treatment Options for Achalasia and Other Esophageal Motility Disorders
Brief Title: Per Oral Endoscopic Myotomy (POEM) and Prolonged Dilatation (PRD) for Achalasia
Acronym: POETA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Erwin Rieder, Priv. Doz. Dr. Erwin Rieder, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POETA
Record Dates: First submitted 2014-12-08; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Per oral endoscopic therapy A (Active Comparator): Per oral endoscopic myotomy
  Interventions: Procedure: Endoscopic intervention A
- Per oral endoscopic therapy B (Active Comparator): Prolonged dilatation by implantation of large diameter stents.
  Interventions: Procedure: Endoscopic intervention B
- Per oral endoscopic therapy C (Active Comparator): Dilatation
  Interventions: Procedure: Endoscopic intervention C
- Laparoscopic surgery (Active Comparator): Laparoscopic Heller myotomy
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Endoscopic intervention A — POEM: Per oral endoscopic myotomy
  Arms: Per oral endoscopic therapy A
Procedure: Endoscopic intervention B — PRD: Prolonged dilatation by temporary implantation of large diameter stent . Stents are additionally attached to the esophageal wall by different technical options.
  Arms: Per oral endoscopic therapy B
Procedure: Endoscopic intervention C — Endoscopic balloon dilatation
  Arms: Per oral endoscopic therapy C
Procedure: Laparoscopic Surgery — Laparoscopic Heller myotomy
  Arms: Laparoscopic surgery

SUMMARY:
Achalasia is an esophageal motility disorder, which leads to clinical symptoms such as dysphagia, regurgitation, chest pain and consecutive weight loss.

Although conventional treatment such as laparoscopic Heller myotomy (LHM) and balloon dilatation (BD) can provide sufficient symptom relief in many patients, both interventions have their individual drawbacks. Additionally, treatment after failed LHM or BD can be challenging and in few might even lead to esophagectomy.

Per oral endoscopic myotomy (POEM) and prolonged dilatation (PRD) are two novel endoscopically performed therapeutic options for achalasia and other esophageal motility disorders. Both not only appear to provide good results, when performed as initial treatment but also might be an excellent option after e.g failed LHM.

The purpose of this study is to evaluate the long-term efficacy of four different treatment options, such as POEM, PRD with stent-fixation, PD and conventional LHM for achalasia in an individualized treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of achalsia, hypertensive lower esophageal sphincter, nutcracker esophagus, or diffuse esophageal spasm

Exclusion Criteria:

* Contraindication for EGD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Achalasia specific symptoms according to the Eckardt score (0-12) | 6 mo post-op
  Eckardt score: Weight loss 0kg (0), less than 5kg (1), 5-10 kg (2), more than 10 kg (3); Dysphagia none(0), occasional (1), daily (2), every meal (3); Regurgitation none(0), occasional (1), daily (2), every meal (3); Retrosternal pain none(0), occasional (1), daily (2), every meal (3)

SECONDARY OUTCOMES:
Barium column height (cm) in esophagogram | 6 mo post-op
Resting pressure (mmHg) at the lower esophageal sphincter | 6 mo post-op
Stent migration | p.o. day 1
  Analysis: On the first postoperative day a routine esophagogram will be used to evaluate the appropriate location of the esophageal stent. Early distal stent dislocation/migration into the stomach will be registered.
Percent of time (min)/24h that the pH is less than 4.0 in pH-metry | 6 mo post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Medical University of Vienna, Vienna, Austria